CLINICAL TRIAL: NCT04703660
Title: Immediate and Carry Over Effect of Different Cervical Mobilization Techniques on Rotator Cuff Tendinitis Patients
Brief Title: Effect of Cervical Mobilization on Rotator Cuff Tendinitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noha Elserty (Other)
Responsible Party: Sponsor-Investigator, Noha Elserty, lecturer of physical therapy, Egyptian Chinese University
Organization: Egyptian Chinese University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: interventional
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Rotator Cuff Tendinitis
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): This group will receive antero-posterior cervical mobilization at c5-6 grade III oscillation
  Interventions: Procedure: cervical mobilization
- group B (Active Comparator): This group will receive lateral glide cervical mobilization at c5-6 grade III oscillation
  Interventions: Procedure: cervical mobilization
- group C (Active Comparator): This group will receive postero-anterior cervical mobilization at c5-6 grade III oscillation
  Interventions: Procedure: cervical mobilization

INTERVENTIONS:
Procedure: cervical mobilization — 3 types of cervical mobilization at the level of C 5- 6

SUMMARY:
this study aimed to investigate the effect of 3 types of cervical mobilization on the strength of shoulder abductors, external rotators and pain level in patient with rotator cuff tendinitis. the measurement will be made immediately, 10 minutes, and 30 minutes after mobilization

DETAILED DESCRIPTION:
subjects will be allocated according to the inclusion and exclusion criteria from outpatient clinic at El sahel teaching hospital. they will be assigned randomly into 3 groups, each group will receive certain type of cervical mobilization. the outcome measures will be measured before, immediate, 10 minutes, and 30 minutes after treatment

ELIGIBILITY:
Inclusion Criteria:

* patients will be included if they have rotator cuff tendinitis

Exclusion Criteria:

* Patients will be excluded if they had recent neck trauma or acute whiplash disorder ,any intra articular injection in the gleno-humeral joint during last three months, patients with musculoskeletal disorder (any type of fracture), any history of surgery on that shoulder and tendon calcification, cervical rib, rotator cuff tear.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
change in strength of shoulder abductors | before treatment, immediate, 10 minutes, and 30 minutes after cervical mobilization
  strength testing with a hand-held dynamometer will be applied for 3 groups using Isometric contraction of shoulder abductors
change in strength of shoulder external rotators | before treatment, immediate, 10 minutes, and 30 minutes after cervical mobilization
  strength testing with a hand-held dynamometer will be applied for 3 groups using Isometric contraction of shoulder external rotators
change in pain level | before treatment, immediate, 10 minutes, and 30 minutes after cervical mobilization
  pain severity will be measured using visual analogue scale for 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Noha S Elserty, PhD, Principal Investigator — Lecturer of physical therapy- Egyptian Chinese University
Locations (1):
- Noha Elserty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
supporting information that will be shared after publication of the study
Supporting Information: Study Protocol, SAP
Time Frame: after publishing the study